CLINICAL TRIAL: NCT03409549
Title: Multi-parametric MRI/Fluorine-18 Fluciclovine PET-CT in Glioblastoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: RD17/101925
Record Dates: First submitted 2018-01-18; First posted 2018-01-24 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Tumor, Brain
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Fluciclovine PET/CT — Fluorine-18 Fluciclovine PET/CT scan of the brain

SUMMARY:
Glioblastoma is the most common adult brain tumour with approximately 2000 new cases each year in the UK.

Optimal treatment consists of surgery followed by radiotherapy and chemotherapy but despite this survival is poor with only 10% of patients alive at 5 years.

Standard imaging (MRI and CT) may not detect the full extent of tumours before treatment and it can be difficult to assess how the tumour is responding to treatment.

The study aims to evaluate more advanced imaging techniques to see if they are better at mapping the whole tumour and assessing response to treatment. Two different imaging techniques will be assessed: Positron Emission Tomography - Computed Tomography (PET-CT) uses a mildly radioactive compound injected into the patient which is taken up into brain tumour cells and shows up as a bright spot on scans. Brain tumours affect blood supply and how much fluid is in the brain tissue as well as how freely fluid can move around. Advanced MR imaging known as multiparametric MRI will be used to look at these additional features. This extra information may help improve planning of radiotherapy and assessing how tumours respond to treatment. Twelve adult patients with glioblastoma undergoing radical treatment will be recruited over a 12 month period. Each patient will have standard MR imaging before radiotherapy (after surgery) and 4-6 weeks following completion of radiotherapy. They will also have advanced MRI and PET/CT before, during and after treatment.

The aim will be to study if this is feasible and could potentially improve radiotherapy planning and response assessment. Imaging will be interpreted by both imaging and brain tumour treatment experts.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* WHO Performance status 0-2 (Appendix 1)
* Histologically proven GBM (WHO Grade 4)
* Clinical decision made to proceed with radical treatment with surgery and chemo-radiotherapy
* Residual tumour following surgery as defined by the surgeons at the time of resection
* Able to provide fully informed written consent
* Able to lie flat for 1 hour
* Not be pregnant or breast feeding. Female patients of childbearing potential must agree to use effective contraception, be surgically sterile, or be post-menopausal.

Exclusion Criteria:

Patients with any of the following are not eligible for the study:

1. Hypersensitivity to Fluorine-18 Fluciclovine
2. Hypersensitivity to MRI contrast media
3. Acute renal failure or moderate renal impairment (estimated glomerular filtration rate < 30 mL/min)
4. Claustrophobia precluding imaging
5. Non-MRI compatible implantable device e.g. pacemaker
6. Uncontrolled pain
7. Urinary incontinence
8. Female patients must not be pregnant and if of child bearing age using adequate contraception
9. Breast feeding
10. Serious psychiatric co-morbidity

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Twelve adult patients with glioblastoma undergoing radical treatment will be recruited
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-10-31 (Estimated); Study Completion 2020-10-31 (Estimated)

PRIMARY OUTCOMES:
Measurment od tumour volumes following scans | 6 months
  The patients tumour volumes from conventional MR, advanced MR and PET/CT will be the primary outcome measure.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nuclear Medicine, St James's University Hospitals, Leeds, United Kingdom

REFERENCES:
- [Derived] Kotecha R, Aboian M, Nabavizadeh SA, Parent EE, Trifiletti DM, Chao ST. Letter regarding "Contribution of PET imaging to radiotherapy planning and monitoring in glioma patients-a report of the PET/RANO group": 18F-fluciclovine and target volume delineation. Neuro Oncol. 2021 Aug 2;23(8):1408-1409. doi: 10.1093/neuonc/noab097. No abstract available. PMID 34081125